CLINICAL TRIAL: NCT04428216
Title: The Efficacy of Ultrasound-Guided Rhomboid Intercostal Block for Pain Management Following Video Assisted Thoracic Surgery
Brief Title: Rhomboid Intercostal Block for Video Assisted Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Primary researcher, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Medipol Hospital 13
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Lung Diseases
Keywords: Video Assisted Thoracic Surgery; Postoperative pain management; Rhomboid intercostal block
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Intervention Model Description: There are two models for this study. The first group is rhomboid intercostal block group. The second one is no intervention control group
Who Masked: Outcomes Assessor
Masking Description: The anesthesiologist who performs postoperative pain evaluation will not know the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group RIB = Rhomboid intercostal block group (Active Comparator): In group RIB, RIB block will be performed with patients in the lateral decubitus position. The linear high frequency probe will be placed in sagittal plane medially on the medial border of the scapula at T5-6 level. The trapezius muscle, rhomboid major muscle, intercostal muscle, ribs and the pleura will be visualized. The needle will be inserted into the fascial plane between the rhomboid major and intercostal muscles in a cranio-caudal direction. A dose of 20 ml 0,25% bupivacaine will be injected into the fascial plane.
  Interventions: Other: Group RIB
- Group C = Control group (No Intervention): Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period. A patient controlled device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol included 10 mcg bolus without infusion dose, 10 min lockout time and 4 hour limit.

INTERVENTIONS:
Other: Group RIB — In group RIB, RIB block will be performed. Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period. A patient controlled device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol included 10 mcg bolus without infusion dose, 10 min lockout time and 4 hour limit.
  Arms: Group RIB = Rhomboid intercostal block group

SUMMARY:
Video assisted thoracic surgery (VATS) has recently been evaluated as the standard surgical procedure for lung surgery. Analgesia management is very important for these patients in postoperative period since insufficient analgesia can cause pulmonary complications such as atelectasis, pneumonia and increased oxygen consumption.

Rhomboid intercostal block (RIB) is a novel block and was first described by Elsharkawy et al. It has been reported that RIB may provide effective analgesia management for several surgeries like thoracotomy.

DETAILED DESCRIPTION:
Following Video Assisted Thoracic Surgery Video assisted thoracic surgery (VATS) has recently been evaluated as the standard surgical procedure for lung surgery. The advantages of VATS prodecures compared with open thoracotomy are rapid recovery, short hospital stay and low complication risk. Although VATS is less painful than thoracotomy, patients may feel severe pain during the first hours at postoperative period. Analgesia management is very important for these patients in postoperative period since insufficient analgesia can cause pulmonary complications such as atelectasis, pneumonia and increased oxygen consumption.

Rhomboid intercostal block (RIB) is a novel block and was first described by Elsharkawy et al. Local anesthetic solution is administrated between the rhomboid muscle and intercostal muscles over the T5-6 ribs 2-3 cm medially of the medial border of the scapula. RIB targets both the posterior rami and lateral cutaneous branches of the thoracic nerves and provides analgesia for the hemithorax from T2 to T9. It has been reported that RIB may provide effective analgesia management for several surgeries like thoracotomy.

The aim of this study is to evaluate the efficacy US-guided Rhomboid intercostal block compared to no intervention control group for postoperative analgesia management after VATS. The primary aim is to compare postoperative opioid consumption and the secondary aim is to evaluate postoperative pain scores (VAS), adverse effects related with opioids (allergic reaction, nausea, vomiting) and complications due to block (pneumothorax, hematoma etc).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for VATS under general anesthesia

Exclusion Criteria:

* history of bleeding diathesis,
* receiving anticoagulant treatment,
* known local anesthetics and opioid allergy,
* infection of the skin at the site of the needle puncture,
* pregnancy or lactation,
* patients who do not accept the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | Change from baseline opioid consumption at postoperative 1, 2, 4, 8, 16, 24 and 48 hours
  The primary aim is to compare perioperative and postoperative opioid consumption

SECONDARY OUTCOMES:
Pain scores (Visual analogue scores-VAS) | Changes from baseline pain scores at postoperative 1, 2, 4, 8, 16, 24 and 48 hours.
  Postoperative pain assessment will be performed using the VAS score (0 = no pain, 10 = the most severe pain felt). The VAS scores at rest and during cough will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will not plan to share IPD

REFERENCES:
- [Background] Elsharkawy H, Saifullah T, Kolli S, Drake R. Rhomboid intercostal block. Anaesthesia. 2016 Jul;71(7):856-7. doi: 10.1111/anae.13498. No abstract available. PMID 27291611
- [Background] Altiparmak B, Korkmaz Toker M, Uysal AI, Turan M, Gumus Demirbilek S. The usage of single-shot ultrasound guided rhomboid intercostal block for analgesia after thoracotomy: Clinical experience in two patients. J Clin Anesth. 2019 Sep;56:98-99. doi: 10.1016/j.jclinane.2019.01.032. Epub 2019 Jan 29. No abstract available. PMID 30708149
- [Background] Yayik AM, Ahiskalioglu A, Ates I, Ahiskalioglu EO, Cinal H. Ultrasound guided bilateral rhomboid intercostal block for breast reduction surgery. J Clin Anesth. 2019 Nov;57:38-39. doi: 10.1016/j.jclinane.2019.03.001. Epub 2019 Mar 6. No abstract available. PMID 30851503